CLINICAL TRIAL: NCT01528020
Title: Treatment of Suicidal and Self-Injurious Adolescents With Emotional Dysregulation
Brief Title: Collaborative Adolescent Research on Emotions and Suicide
Acronym: CARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other); University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Marsha Linehan, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41565-C; R01MH090159-01A1 (NIH)
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Suicidal and Self-injurious Behaviour
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dialectical Behavior Therapy (Experimental)
  Interventions: Behavioral: Dialectical Behavior Therapy
- Inidividual and Group Supportive Therapy (Active Comparator)
  Interventions: Behavioral: Individual and Group Supportive Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — DBT is a cognitive behavioral approach to treatment that synthesizes change based strategies characteristic of behavior therapy and validation strategies consistent with acceptance based treatments through application of dialectical principles and techniques. Based on a combined capability deficit and motivational model which states that 1) adolescents with suicidal behaviors and borderline features lack important interpersonal, self-regulation and distress tolerance skills, and 2) personal and environmental factors often both block and/or inhibit use of behavioral skills that adolescents do have, and at times reinforce dysfunctional behaviors. The primary adaptation for adolescents is the inclusion of family in the DBT skills training portion of therapy as well as a much greater inclusion of parents in the management of high suicide risk.
  Arms: Dialectical Behavior Therapy
Behavioral: Individual and Group Supportive Therapy — The aim of IGST is relief or reduction of symptoms, the promotion of personal growth including enhancement of adolescents' strengths/coping skills and capacity to use environmental supports and to help suicidal adolescents increase their sense of self-esteem. Treatment aims to reduce suicidal behavior and emotion dysregulation by helping the adolescent learn to trust and validate themselves. The overarching assumption in IGST is that adolescents become suicidal for a variety of reasons, but they often report feeling isolated, misunderstood, unloved and unwanted. IGST Interventions include providing a strong therapeutic alliance where the therapist provides an environment that is completely trusting and validating to counter the experience of the depressed/suicidal youth.
  Arms: Inidividual and Group Supportive Therapy

SUMMARY:
Suicide is the third leading cause of death among adolescents in the US yet there is a paucity of research on effective treatments for this population. The primary aim of the research described in this application is to evaluate the efficacy of dialectical behavior therapy (DBT) for suicidal adolescents. DBT has an empirical track record with suicidal adults of reducing the incidence, frequency and medical risk of suicide attempts and non-suicidal self-injuries among individuals meeting criteria for borderline personality disorder (BPD). While DBT is widely used in the community with suicidal adolescents, particularly those with difficulties characteristic of BPD such as poor emotion regulation and impulse control, no randomized trial of DBT with suicidal adolescents has ever been conducted. And, while non-randomized trials indicate that the intervention is both safe and effective, without a randomized trial the investigators simply do not know whether DBT for suicidal adolescents is efficacious or not. Given the severity of the problem and the lack of alternative treatments for high risk adolescents, addressing this question is of great importance. The second aim of the research is to analyze mediators of reduced suicidal and self-injurious behaviors in adolescents. 170 adolescents at two sites (Seattle and Los Angeles) will be randomized to DBT or Individual and Supportive Group Therapy (IGST). Both treatments include 6 months of individual and group treatment and adolescents and a parent complete 5 assessments over a 1-year period.

ELIGIBILITY:
Inclusion Criteria:

1. Current suicide ideation;
2. More than one intentional self-injury or suicide attempt;
3. Has difficulties with emotion and impulsive behavior or has characteristics similar to borderline personality disorder;
4. 13-17 years of age;
5. At least one family member or responsible adult available to participate in assessments and treatment.

Exclusion Criteria:

* Has significant developmental delays
* Has significant current mania, psychosis or life threatening anorexia
* Has a court order for treatment

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2012-01; Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Suicide Events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marsha M Linehan, Ph.D., Principal Investigator — University of Washington; Elizabeth A McCauley, Ph.D., Principal Investigator — Seattle Children's Hospital; Joan Asarnow, Principal Investigator — University of California, Los Angeles; Michele Berk, Ph.D., Principal Investigator — Harbor UCLA
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Derived] Berk MS, Gallop R, Asarnow JR, Adrian MC, Hughes JL, McCauley E. Remission, Recovery, Relapse, and Recurrence Rates for Suicide Attempts and Nonsuicidal Self-Injury for Suicidal Youth Treated With Dialectical Behavior Therapy or Supportive Therapy. J Am Acad Child Adolesc Psychiatry. 2024 Sep;63(9):888-897. doi: 10.1016/j.jaac.2024.01.012. Epub 2024 Feb 5. PMID 38325518
- [Derived] Berk MS, Gallop R, Asarnow JR, Adrian M, Avina C, Hughes JL, Korslund KE, McCauley E. Trajectories of Treatment Response and Nonresponse in Youth at High Risk for Suicide. J Am Acad Child Adolesc Psychiatry. 2022 Sep;61(9):1119-1130. doi: 10.1016/j.jaac.2022.01.010. Epub 2022 Feb 2. PMID 35122952
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] Asarnow JR, Berk MS, Bedics J, Adrian M, Gallop R, Cohen J, Korslund K, Hughes J, Avina C, Linehan MM, McCauley E. Dialectical Behavior Therapy for Suicidal Self-Harming Youth: Emotion Regulation, Mechanisms, and Mediators. J Am Acad Child Adolesc Psychiatry. 2021 Sep;60(9):1105-1115.e4. doi: 10.1016/j.jaac.2021.01.016. Epub 2021 Feb 1. PMID 33539915
- [Derived] McCauley E, Berk MS, Asarnow JR, Adrian M, Cohen J, Korslund K, Avina C, Hughes J, Harned M, Gallop R, Linehan MM. Efficacy of Dialectical Behavior Therapy for Adolescents at High Risk for Suicide: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Aug 1;75(8):777-785. doi: 10.1001/jamapsychiatry.2018.1109. PMID 29926087
- See also: Related Info — http://depts.washington.edu/brtc/
- See also: Related Info — http://www.harboruclapsych.com